CLINICAL TRIAL: NCT06165770
Title: Cornual Pregnancy: Results of a Single-center Retrospective Experience and Systematic Review on Reproductive Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, Principal investigator, University of Palermo
Other Study IDs: CORNUAL_pregnancies
Record Dates: First submitted 2023-11-18; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Ectopic Pregnancy
Keywords: cornual pregnancy; ectopic pregnancy; laparoscopy; methotrexate; fertility
MeSH Terms: conditions — Pregnancy, Ectopic; Pregnancy, Cornual | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopy — Conservative or surgery treatment for cornual pregnancies

SUMMARY:
To present our experience in the diagnosis and management of cornual pregnancy. A systematic review was also conducted to investigate reproductive outcomes after treatment.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* patients with a diagnosis of cornual pregnancies.

Exclusion Criteria:

* All patients whose medical records did not contain the data deemed necessary for study analysis or who did not consent to the publication and use of their data;
* Other type of ectopic pregnancies.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Patients with a diagnosis of Cornual pregnancy aged ≥ 18.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 2 years
  defined as the presence of a gestational sac on transvaginal ultrasound or other definitive clinical signs
ongoing pregnancy rate | 2 years
  defined as a pregnancy beyond 24 weeks of gestation
miscarriage rate | 2 years
  defined as fetal loss before the 20th week of gestation